CLINICAL TRIAL: NCT05213923
Title: ED Tracking Sheet Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Harman S. Gill, Principal Investigator, Assistant Professor of Emergency Medicine and Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001224
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Sepsis; Severe Sepsis; Systemic Inflammatory Response Syndrome
Keywords: CMS Compliance; ED Pharmacist
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention (No Intervention): Patients presenting to the Emergency Department meeting severe sepsis criteria prior to implementation of an ED Sepsis Tracking Sheet
- Post-intervention (Experimental): Patients presenting to the Emergency Department meeting severe sepsis criteria following implementation of an ED Sepsis Tracking Sheet
  Interventions: Procedure: ED Sepsis Tracking Sheet

INTERVENTIONS:
Procedure: ED Sepsis Tracking Sheet — Implementation of an ED Sepsis Tracking Sheet. This sheet will track time of patient presentation, time of High-Acuity Medical Response (HAMR) page, time of bilateral 18g or larger IV access, time of initial lactate, time two sets of blood cultures were sent, time antibiotics were administered as well as which antibiotics and what dose, time initial IV fluid bolus was completed, time repeat lactate was sent, timing of post-IV-fluid bolus vital signs, as well as the presence of persistent hypotension following this IV fluid bolus and whether or not vasopressors were applied.
  Arms: Post-intervention

SUMMARY:
The purpose of this study is to assess whether implementation of an ED Sepsis Tracking Sheet effects the percentage of goal-directed sepsis criteria met in a tertiary care academic Emergency Department.

DETAILED DESCRIPTION:
Sepsis remains a common cause of morbidity and mortality in the hospital setting. Accurate diagnosis and timely initiation of therapy are important drivers of patient-centered outcomes in sepsis management. Compliance with the core measures listed in the surviving sepsis campaign guidelines has been variable.

An ED-specific Sepsis Tracking Sheet (STS) - a tool for implementing and documenting critical actions in sepsis management - was created at our institution by a team of physicians, nurses, and ED pharmacists. Dedicated ED pharmacists were instructed to fill this sheet within one hour of the sepsis-specific best practice advisory (BPA) being activated in the ED. Core measures associated with the one hour and three hour sepsis bundles were tracked and outcomes were compared pre- and post-implementation of the STS.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Initially evaluated in the DHMC Lebanon Emergency Department
* Activated sepsis BPA upon initial presentation (triage history consistent with infection combined with 2 or more SIRS criteria? Are these the criteria that trigger our sepsis BPA?)

Exclusion Criteria:

* Patients who are transferred to the DHMC Lebanon Emergency Department from another facility
* Patients with absent data regarding one or more of the goal-directed sepsis criteria
* Patients who did not initially meet criteria to trigger the sepsis BPA, but developed sepsis later in their hospital course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of goal-directed sepsis criteria met | Time of ED presentation to the time of in-hospital death or hospital discharge, approximately 2 weeks
  Goal-directed sepsis criteria involve the following: 1) Was an initial lactate obtained? 2) Were two sets of blood cultures sent? 3) Were antibiotics given within one hour of identification of severe sepsis? 4) Was the patient given an initial IV fluid bolus? 5) Was a repeat lactate sent if the initial lactate was elevated? These five criteria will be assessed as "met" or "not met" for each patient. The total of "met" and "not met" criteria will be aggregated across patients. The percentage of goal-directed sepsis criteria met will be calculated as "met" criteria divided by the sum of "met" plus "not met" criteria.

SECONDARY OUTCOMES:
Length of hospital stay | Time of ED presentation to the time of in-hospital death or hospital discharge, approximately 2 weeks
  Time of ED presentation to the time of in-hospital death or hospital discharge, measured in days.
In-hospital mortality | Time of ED presentation to the time of in-hospital death or hospital discharge, approximately 2 weeks
  Death attributed to any cause occurring at any time between the patient's ED presentation and hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Harman Gill, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans for sharing IPD at this time.

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Mayr FB, Yende S, Angus DC. Epidemiology of severe sepsis. Virulence. 2014 Jan 1;5(1):4-11. doi: 10.4161/viru.27372. Epub 2013 Dec 11. PMID 24335434
- [Background] Levy MM, Rhodes A, Phillips GS, Townsend SR, Schorr CA, Beale R, Osborn T, Lemeshow S, Chiche JD, Artigas A, Dellinger RP. Surviving Sepsis Campaign: association between performance metrics and outcomes in a 7.5-year study. Crit Care Med. 2015 Jan;43(1):3-12. doi: 10.1097/CCM.0000000000000723. PMID 25275252
- [Background] Coba V, Whitmill M, Mooney R, Horst HM, Brandt MM, Digiovine B, Mlynarek M, McLellan B, Boleski G, Yang J, Conway W, Jordan J; (The Henry Ford Hospital Sepsis Collaborative Group). Resuscitation bundle compliance in severe sepsis and septic shock: improves survival, is better late than never. J Intensive Care Med. 2011 Sep-Oct;26(5):304-13. doi: 10.1177/0885066610392499. Epub 2011 Jan 10. PMID 21220270
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Fleischmann-Struzek C, Mellhammar L, Rose N, Cassini A, Rudd KE, Schlattmann P, Allegranzi B, Reinhart K. Incidence and mortality of hospital- and ICU-treated sepsis: results from an updated and expanded systematic review and meta-analysis. Intensive Care Med. 2020 Aug;46(8):1552-1562. doi: 10.1007/s00134-020-06151-x. Epub 2020 Jun 22. PMID 32572531
- [Background] Schorr C, Odden A, Evans L, Escobar GJ, Gandhi S, Townsend S, Levy M. Implementation of a multicenter performance improvement program for early detection and treatment of severe sepsis in general medical-surgical wards. J Hosp Med. 2016 Nov;11 Suppl 1:S32-S39. doi: 10.1002/jhm.2656. PMID 27805796
- [Background] Downing NL, Rolnick J, Poole SF, Hall E, Wessels AJ, Heidenreich P, Shieh L. Electronic health record-based clinical decision support alert for severe sepsis: a randomised evaluation. BMJ Qual Saf. 2019 Sep;28(9):762-768. doi: 10.1136/bmjqs-2018-008765. Epub 2019 Mar 14. PMID 30872387